CLINICAL TRIAL: NCT01598870
Title: Redefinition of Diagnostic Criteria for Spontaneous Bacterial Peritonitis: Assessment of Accuracy of Available Tests and of Reference Standard
Brief Title: Diagnosis of Spontaneous Bacterial Peritonitis
Acronym: ARSDIASP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Lecco (Other)
Responsible Party: Principal Investigator, Agostino Colli, MD, Head of Internal Medicine Department AO Provincia di Lecco, Azienda Ospedaliera di Lecco
Other Study IDs: AOLecco001
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Spontaneous Bacterial Peritonitis
Keywords: Spontaneous bacterial peritonitis.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and ascitic fluid samples stored at -80°C
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with cirrhosis and ascites: Patients requiring diagnostic and/or therapeutic paracentesis.
  Interventions: Other: Diagnostic tests

INTERVENTIONS:
Other: Diagnostic tests — Leukocyte count by automated counters; reagent strips for leukocyte esterase and for lactoferrin; ascitic fluid pH; leukocyte cytometry; bacterial DNA detection and quantification.

SUMMARY:
The study is aimed to revise the current criteria for the diagnosis of spontaneous bacterial peritonitis and the decisional thresholds to start treatment. The accuracy of current diagnostic tests will be compared with that of new tests, which could potentially become more accurate reference standards. This could lead to the definition of a more accurate and effective diagnostic algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis and ascites with clinical indication to carry out a diagnostic and/or therapeutic paracentesis.

Exclusion Criteria:

* Etiology of ascites other than cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis and ascites requiring paracentesis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-07 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Comparing the accuracy of current reference standard for the diagnosis of spontaneous bacterial peritonitis, i.e. neutrophil count in ascitic fluid of >250/mm3 as determined by microscopy, with alternative diagnostic tests. | One month
  Reference standard is neutrophil count in ascitic fluid of >250/mm3 as determined by microscopy.
  Alternative diagnostic tests are: Leukocyte count by automated counters; reagent strips for leukocyte esterase and for lactoferrin; ascitic fluid pH; leukocyte cytometry; bacterial DNA detection and quantification.
  Discrepancies between reference standard and alternative tests will be assessed by one month clinical follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Agostino Colli, MD, Principal Investigator — AO Provincia di Lecco, Department of Medicine, A. Manzoni Hospital, Lecco
Locations (1):
- Department of Medicine, A. Manzoni Hospital, Lecco, Italy